CLINICAL TRIAL: NCT01847833
Title: Advanced MRI Applications Development
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Elizabeth R. Gerstner, MD, Dr., Massachusetts General Hospital
Other Study IDs: 2012p001007
Record Dates: First submitted 2013-01-11; First posted 2013-05-07 (Estimated); Last update posted 2018-03-26 (Actual); Status verified 2018-03

CONDITIONS: Brain Tumors
MeSH Terms: conditions — Brain Neoplasms | interventions — Magnetic Resonance Spectroscopy

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Patients with brain tumors
  Interventions: Other: MRI scan

INTERVENTIONS:
Other: MRI scan

SUMMARY:
The goals of this study are to:

1. To improve upon and develop new innovative magnetic resonance imaging techniques that refine image quality and enhance performance. Improvements in these areas will have positive implications for medical diagnosis and treatment.
2. To correlate MRI images with underlying disease pathophysiology in order to ensure that imaging accurately reflects the disease process.

ELIGIBILITY:
Inclusion Criteria:

* Brain Tumor

Exclusion Criteria:

* Unable to undergo MRI

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients with brain tumors or tumors affecting the brain.
Sampling Method: Non-Probability Sample
Dates: Start 2014-01; Primary Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
patients alive and progression free at 6 months | 6 months

CONTACTS AND LOCATIONS:
Locations (1):
- MGH, Boston, Massachusetts, United States